CLINICAL TRIAL: NCT05516979
Title: A Double-blind, Multi-center, Randomized, Placebo-controlled Study of the Safety and Efficacy of 12 Weeks Extended Treatment With AP1189 in Early Rheumatoid Arthritis (RA) Patients naïve to DMARD Treatment
Brief Title: A Safety & Efficacy Study of Treatment With AP1189 in Rheumatoid Arthritis Patients naïve to DMARD Treatment
Acronym: EXPAND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SynAct Pharma Aps (Industry)
Collaborators: NBCD A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SynAct-CS007
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — N-(3-(1-(2-nitrophenyl)-1H-pyrrol-2-yl)allylidenamino)guanidine

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized, double-blind, placebo-controlled study with 12 weeks of treatment with AP1189 or placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 100 mg AP1189 (Experimental): Treatment period of 12 weeks given as 1 tablet daily
  Interventions: Drug: 100 mg AP1189
- Placebo (Placebo Comparator): Treatment period of 12 weeks given as 1 tablet daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 100 mg AP1189 — AP1189 tablets for oral use
  Other Names: AP1189 tablets for oral use
  Arms: 100 mg AP1189
Drug: Placebo — Matching placebo for oral use
  Arms: Placebo

SUMMARY:
The study is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of 12 weeks daily treatment with 100 mg AP1189 in RA patients who are to start up-titration with methotrexate (MTX).

ELIGIBILITY:
Main Inclusion Criteria:

* Confirmed diagnosis of RA according to the 2010 ACR/EULAR RA classification criteria and are ACR class I-III
* ≥ 6 swollen joints (based on 66 joint counts) and ≥ 6 tender joints (based on 68 joint counts).
* Candidate for MTX treatment
* Is about to begin treatment with MTX
* Must meet at least one of the following parameters at Screening:

  1. positive result for anti-CCP or RF
  2. Serum CRP ≥ 6 mg/L
* Highly active RA (CDAI > 22) at screening and baseline
* Negative QuantiFERON-in-Tube test (QFG-IT)
* Females of child-bearing potential must use of highly effective birth control method

Main Exclusion Criteria:

* Major surgery (including joint operation) within 8 weeks prior to screening or planned surgery within 1 month following randomization
* Rheumatic autoimmune disease other than RA, including systemic lupus erythematosus (SLE), mixed connective tissue disease (MCTD), scleroderma, polymyositis, or significant systemic involvement secondary to RA. Sjögren's syndrome with RA is allowable
* Prior history of or current inflammatory joint disease other than RA
* Subjects with fibromyalgia
* Use of hydroxychloroquine within 4 weeks prior the Screening Visit
* Initiation of, or change in existing NSAID treatment within 2 weeks prior to the baseline visit
* Corticosteroids except inhaled or nasal formulations for seasonal allergy or asthma are prohibited within 2 weeks prior to screening
* Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary, renal, hepatic, endocrine, or gastrointestinal disease
* Have prior renal transplant, current renal dialysis, or severe renal insufficiency
* Uncontrolled disease states, such as asthma, psoriasis, or inflammatory bowel disease where flares are commonly treated with oral or parenteral corticosteroids
* Evidence of active malignant disease (except basal cell carcinoma of the skin that has been excised and cured)
* Neuropathies or other painful conditions that might interfere with pain evaluation
* Body weight of >150 kg
* HBsAg positive and/or Anti-HBc with sign of current infection.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Number of reported AEs | 12 weeks
  Evaluation of the safety and tolerability of AP1189 on the number and severity of reported Adverse Events, compared with placebo
Change in ACR20 | 12 weeks
  The change in American College of Rheumatology 20% (ACR20) compared to baseline

SECONDARY OUTCOMES:
Change in ACR50 | 12 weeks
  The change in American College of Rheumatology 50% (ACR50) compared to baseline
Change in ACR70 | 12 weeks
  The change in American College of Rheumatology 70% (ACR70) compared to baseline
Change in (CDAI) | 12 weeks
  The change Clinical Disease Activity Index (CDAI) compared to baseline
Change in DAS-28 | 12 weeks
  The change in DAS-28, based on a CRP value, compare to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Timofei Mosneaga Republican Clinical Hospital, Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: No